CLINICAL TRIAL: NCT06527404
Title: A Phase 3, 52-Week, Multicenter, Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy, Safety, and Tolerability of Rocatinlimab in Adult Subjects With Prurigo Nodularis Who Are Inadequately Controlled on Topical Therapies or Not Eligible for Topical Therapies
Brief Title: A Phase 3, Placebo-controlled, Double-blind Study Assessing Rocatinlimab in Prurigo Nodularis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230053
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prurigo Nodularis
Keywords: Rocatinlimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Blinded Treatment (Experimental): Participants will receive rocatinlimab dose 1 subcutaneously (SC) during Treatment Period A and B.
  Interventions: Drug: Rocatinlimab
- Arm B: Blinded Treatment (Experimental): Participants will receive rocatinlimab dose 2 SC during Treatment Period A and B.
  Interventions: Drug: Rocatinlimab
- Arm C: Blinded Treatment (Experimental): Participants will receive matching placebo SC during Treatment Period A and B.
  Interventions: Drug: Placebo
- Arm D: Open-label (Experimental): Participants will receive open-label rocatinlimab dose 1 SC during Treatment Period B.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — SC Injection
  Other Names: AMG 451
  Arms: Arm A: Blinded Treatment; Arm B: Blinded Treatment; Arm D: Open-label
Drug: Placebo — SC Injection
  Arms: Arm C: Blinded Treatment

SUMMARY:
The main objective of the study will be to evaluate the efficacy of rocatinlimab compared with placebo at week 24 on the patient-reported outcome (PRO) measure of pruritus and overall clinical assessment score (US only).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (or any legal adult age within the country if it is older than 18 years)
* Clinical Diagnosis of Prurigo Nodularis that has been present for at least 3 months.
* Patient-reported average Daily Itch Score based on electronic daily diary assessment the last 7 days prior to and including day 1.
* Has ≥ 20 prurigo nodularis nodules in total with bilateral distribution on both legs and /or arms and /or trunk.
* History of inadequate response to topical therapies of medium or higher potency or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks).

Exclusion Criteria:

* Skin or systemic morbidities, other than prurigo nodularis, that have been active within the last 3 months that interfere with assessment of study outcomes including but not limited to atopic dermatitis (signs or symptoms other than dry skin or requiring treatment is not allowed; use of emollients and/or history of AD is allowed).
* Prurigo nodularis secondary to medications.
* Prurigo nodularis secondary to neurologic or psychiatric medical conditions.
* Treatment with any systemic biologic immunosuppressive or systemic biologic immunomodulatory therapy for prurigo nodularis or any other autoimmune, inflammatory, or allergic disease within 12 weeks or 5 half-lives, whichever is longer, prior to day 1 prerandomization.
* Treatment with live virus including live attenuated vaccination 12 weeks prior to day 1 prerandomization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Global: Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score at Week 24 | Up to 24 weeks
US Only: Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score and Prurigo Nodularis Stage Assessment at Week 24 | Up to 24 weeks

SECONDARY OUTCOMES:
Global: Number of Participants Achieving Improvement in Prurigo Nodularis Stage Assessment Score at Week 24 | Week 24
Global: Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score and Prurigo Nodularis Stage Assessment at Week 24 | Baseline and Week 24
Global: Percentage Improvement from Baseline in Weekly Average of Daily Itch Score at Week 24 | Baseline and Week 24
Global: Number of Participants Achieving Reduction in Weekly Average Daily Prurigo Nodularis Skin Pain Assessment at Week 24 in Those with Baseline NRS Above Cutoff | Baseline and Week 24
US Only: Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score at Week 24 | Baseline and Week 24
US Only: Number of Participants with Improvement in Prurigo Nodularis Stage Assessment at Week 24 | Week 24
US Only: Percent Improvement from Baseline in Weekly Average of Daily Itch Score at Week 24 | Week 24
US Only: Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Skin Pain Assessment at Week 24 in Participants With Baseline Score Greater Than or Equal to a Cutoff Score | Week 24
Change from Baseline in Weekly Average of Daily Itch Score at Weeks 24, 36 and 52 | Baseline, Week 24, Week 36 and Week 52
Percent Improvement from Baseline in Weekly Average of Daily Itch Score at Week 36 and 52 | Baseline, Week 36 and Week 52
Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score at Weeks 16, 36 and 52 | Baseline, Week 16, Week 36 and Week 52
Number of Participants Achieving Weekly Average of Daily Itch Score Less than a Cutoff Score at Week 36 and 52 | Week 36 and Week 52
Change from Baseline in Prurigo Nodularis Stage Assessment Score at Week 24, 36, and 52 | Baseline, Week 24, Week 36 and Week 52
Number of Participants Achieving Improvement in Prurigo Nodularis Stage Assessment Score at Weeks 36 and 52 | Week 36 and Week 52
Number of Participants Achieving Improvement in Prurigo Nodularis Activity Assessment Score at Weeks 24, 36 and 52 | Week 24, Week 36 and Week 52
Change from Baseline in Quality of Life Assessment Score at Weeks 24, 36 and 52 | Baseline, Week 24, Week 36 and Week 52
Number of Participants Achieving Reduction from Baseline in Quality of Life Assessment Score at Weeks 24, 36 and 52 in Participants with Baseline Score Greater Than or Equal to a Cutoff Score | Baseline, Week 24, Week 36 and Week 52
Change from Baseline in Weekly Average of Daily Skin Pain Assessment Score at Weeks 24, 36 and 52 | Baseline, Week 24, Week 36 and Week 52
Change from Baseline in Weekly Average of Daily Sleep Disturbance Assessment Score at Weeks 24, 36 and 52 | Baseline, Week 24, Week 36 and Week 52
Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Sleep Disturbance Assessment Score at Weeks 24, 36 and 52 in Participants with Baseline Weekly Average Score Greater Than or Equal to a Cutoff Score | Baseline, Week 24, Week 36 and Week 52
Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Itch Score and Prurigo Nodularis Stage Assessment at Week 36 and 52 | Baseline, Week 36 and Week 52
Number of Participants Achieving Reduction from Baseline in Weekly Average of Daily Skin Pain Assessment Score at Week 36 and 52 in Participants With Baseline Score Greater Than or Equal to a Cutoff Score | Baseline, Week 36 and Week 52
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately Week 68
  An adverse event (AE) is any untoward medical occurrence in a clinical study subject irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration will be recorded as TEAEs. A serious TEAE is any untoward medical occurrence that meets one of the following criteria: Is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or another medically important serious event.
Number of Participants Experiencing AEs of Special Interest (EOIs) | Up to approximately Week 68
Number of Participants with Anti-rocatinlimab Antibodies | Baseline to Week 68
Serum Concentrations of Rocatinlimab | Baseline to Week 52
Trough Concentration (Ctrough) of Rocatinlimab | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (192):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - First OC Dermatology, Fountain Valley, California
  - Los Angeles Universal Research Center, Los Angeles, California
  - Paradigm Clinical Research Center Inc, San Diego, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Southern Clinical Research, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Clinical Research Trials of Florida Inc, Tampa, Florida
  - Olympian Clinical Research - Tampa, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Endeavor Health Clinical Trials Center, Skokie, Illinois
  - The Indiana Clinical Trials Center PC, Plainfield, Indiana
  - Revival Research Institute, LLC, Troy, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Optima Research, Boardman, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Center For Clinical Studies PLLC, Houston, Texas
  - Clarity Dermatology, Lancaster, Texas
  - Springville Dermatology, Springville, Utah
- Argentina (6):
  - Hospital Universitario Austral, Derqui, Pilar, Buenos Aires
  - Instituto de Investigaciones Clinicas de Cordoba, Córdoba, Córdoba Province
  - Instituto de Neumonologia y Dermatologia, Buenos Aires, Distrito Federal
  - Derma Internacional, Buenos Aires, Distrito Federal
  - Centro de investigacion clinica y epidemiologica, San Miguel D Tucuman, Tucumán Province
  - Parra Dermatologia, Mendoza
- Australia (5):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
- Belgium (3):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitaire Ziekenhuizen Leuven Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Brazil (6):
  - Clinica Instituto Bahiano de Imunoterapia - Medicina, Reumatologia e Dermatologia ltda, Salvador, Estado de Bahia
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual Paulista Julio de Mesquita Filho, Botucatu, São Paulo
  - Fundacao Abc - Centro Univ Fmabc, Santo André, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Canada (12):
  - Doctor Chih-Ho Hong Medical Incorporated, Surrey, British Columbia
  - Skincare Studio, St. John's, Newfoundland and Labrador
  - CCA Medical Research Corp, Ajax, Ontario
  - Centricity Research London Victoria, London, Ontario
  - Lovegrove Dermatology, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Toronto Research Centre Inc, Toronto, Ontario
  - AvantDerm, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
- Chile (5):
  - Enroll SpA, Providencia, Santiago Metropolitan
  - Centro Medico Skinmed Spa, Santiago
  - Fundacion Innovacion Cardiovascular Clinica Ensenada, Santiago
  - Centro Internacional de Estudios Clinicos, Santiago
  - Clinical Research Chile SpA, Valdivia
- China (20):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital Sun-Yat Sen University, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital Of Xi An Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Affiliated Hangzhou First Peoples Hospital School of Medicine Westlake University, Hangzhou, Zhejiang
- Finland (3):
  - Clinical Research Services Helsinki, Helsinki
  - Oulun Yliopistollinen sairaala, Oulu
  - Terveystalo Tampere, Tampere
- France (5):
  - Centre Hospitalier Regional Universitaire de Brest - Hopital Morvan, Brest
  - Centre Hospitalier Le Mans, Le Mans
  - Cabinet du Docteur Ruer-Mulard Mireille, Martigues
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Centre Hospitalier Universitaire de Rouen - Hopital Charles Nicolle, Rouen
- Germany (11):
  - Universitaetsklinikum Augsburg, Augsburg
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Rosenpark Research GmbH, Darmstadt
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsmedizin Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Hautarztpraxis Mortazawi, Remscheid
  - Universitaetsklinikum Tuebingen, Tübingen
  - Helios Klinikum Wuppertal, Wuppertal
- Greece (5):
  - University General Hospital Attikon, Athens
  - Andreas Syngros Hospital Of Venereal And Dermatological Diseases, Athens
  - General Hospital Of Nea Ionia Konstantopouleio Patision, Nea Ionia
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital, Thessaloniki
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Hungary (6):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Derm-Surg Kft, Kaposvár
  - DermaMed Research Kft, Orosháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Italy (5):
  - Ospedale San Salvatore, LAquila
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Fondazione Policlinico Tor Vergata, Roma
- Japan (15):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaido
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kawasaki Medical School Hospital, Kurashiki-shi, Okayama-ken
  - Hayami Dermatology Clinic, Osaka, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - National Defense Medical College hospital, Tokorozawa-shi, Saitama
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Tokyo Teishin Hospital, Chiyoda-ku, Tokyo
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
  - Tokyo Medical University Hospital, Shinjyuku-ku
- Latvia (3):
  - J Kisis, Riga
  - Outpatient clinic Veselibas Centrs 4, Riga
  - Outpatient clinic Veselibascentrs 4, Riga
- Mexico (2):
  - Clínica de Enfermedades Crónicas y de Procedimientos Especiales, Morelia, Michoacán
  - Instituto de Investigaciones Aplicadas a la Neurociencia A C, Durango
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (12):
  - Niepubliczny Zaklad Opieki Zdrowotnej, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - AKK Medical Spolka z ograniczona odpowiedzialnoscia Centrum Medyczne Tu sie leczy, Gdansk
  - GynCentrum Spzoo NZOZ Holsamed - Oddzial Libero, Katowice
  - Amicare Spolka z ograniczona odpowiedzialnoscia Spolka Komandytowa Amicare Centrum Medyczne, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Uniwersytecki Szpital Kliniczny imienia Fryderyka Chopina w Rzeszowie, Rzeszów
  - Velocity Skierniewice Spolka z Ograniczona Odpowiedzialnoscia, Skierniewice
  - Centrum Zdrowia Dziecka i Rodziny Im Jana Pawla II w Sosnowcu Osrodek Badan Klinicznych, Sosnowiec
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spolka Partnerska, Wroclaw
  - DermMedica Spzoo Centrum Columbus, Wroclaw
- Portugal (3):
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Hospital Cuf Descobertas, Lisbon
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- South Korea (7):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (8):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (2):
  - Diagnostiskt Centrum Hud i Sickla, Nacka
  - Akademiska sjukhuset, Uppsala
- Switzerland (2):
  - Inselspital Bern, Bern
  - Universitaetsspital Zuerich, Zuerich Flughafen
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (6):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Adnan Menderes Universitesi Medical Faculty, Aydin
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Izmir Demokrasi Universitesi Buca Seyfi Demirsoy Egitim ve Arastirma Hastanesi, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (5):
  - Queen Elizabeth University Hospital, Glasgow
  - Chapel Allerton Hospital, Leeds
  - Royal London Hospital, London
  - Guys Hospital, London
  - Ameli-Biogroup Limited, Waltham Abbey

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com